CLINICAL TRIAL: NCT00464594
Title: A Randomized Comparative Clinical Study on Suppression of Progression From Early Diabetes, Diet/Exercise Standard Intervention vs. Concurrent Pharmacological Standard Intervention
Brief Title: Japan Early Diabetes Intervention Study
Acronym: JEDIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Japan Early Diabetes Intervention Study Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JEDIS ver.4.0; UMIN000000681
Record Dates: First submitted 2007-04-19; First posted 2007-04-23 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: Diabetes Mellitus
Keywords: Japan Early Diabetes Intervention Study
MeSH Terms: conditions — Diabetes Mellitus | interventions — Acarbose; Metformin; Gliclazide

INTERVENTIONS:
Behavioral: Standard lifestyle guidance
Drug: Lifestyle guidance and monotherapy with acarbose
Drug: Lifestyle guidance and monotherapy with metformin
Drug: Lifestyle guidance and monotherapy with gliclazide

SUMMARY:
The purpose of this study is to compare the suppressive effect of two kinds of interventions on the worsening/progression to definite diabetes: standard lifestyle guidance and standard lifestyle guidance combined with pharmacological intervention (monotherapy with one of acarbose, metformin, or gliclazide).

DETAILED DESCRIPTION:
In newly-diagnosed early diabetes patients, a randomized comparative study will be conducted to compare the suppressive effect of the following two kinds of interventions on the worsening/progression to definite diabetes which has a harmful hyperglycemia i.e. an increased risk of microangiopathy: standard education for the improvement of lifestyle in accordance with the "Guidelines for the Treatment of Diabetes Mellitus in Japan" of the Japan Diabetes Society (JDS) and standard lifestyle guidance combined with pharmacological intervention using the lowest possible dose of commercially available oral hypoglycemic agents (one of acarbose, metformin, or gliclazide) in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Results of 75-g oral glucose tolerance test (75 g OGTT)will be used to confirm FPG <= 125 mg/dL, 2-h PG >= 200 mg/dL and HbA1c <= 6.9%

Exclusion Criteria:

* Type 1 diabetes mellitus
* Undergoing treatment with steroids
* Secondary diabetes mellitus
* Diabetes mellitus due to suspected gene abnormalities
* BMI >= 35 kg/m2 or BMI < 18.5 kg/m2
* Undergone a surgery
* Severe hyperuricemia (gout) associated with organ dysfunction
* Severe vascular diseases with organ dysfunction
* Cancer or other malignant neoplasms
* Liver cirrhosis or chronic hepatic, chronic renal failure
* Gastrointestinal disorders
* Always performing rigorous muscular exercise
* Severe infection or serious trauma
* Women who are pregnant
* Alcohol dependence or drug dependence
* Drug allergy
* Anemic
* Abnormal hemoglobinuria
* Severe mental disease

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2560
Dates: Start 2007-04

PRIMARY OUTCOMES:
FPG >= 140mg/dl and HbA1c >= 7.0%

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kuzuya, Principal Investigator — Jichi Medical University
Locations (1):
- Tokyo Medical and Dental University, Tokyo, Japan